CLINICAL TRIAL: NCT01345539
Title: Phase II Study for Curative Intent Treatment for Patients With Oligometastatic Disease at Initial Presentation
Brief Title: Radiosurgery for Patients With Oligometastatic Disease at Initial Presentation
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Participant enrollment was negatively impacted by medical oncology treatment with systemic therapy alone and accrual to other clinical trials.
Sponsor: Steven Burton (Other)
Responsible Party: Sponsor-Investigator, Steven Burton, Clinical Associate Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCC 10-027
Record Dates: First submitted 2011-02-17; First posted 2011-05-02 (Estimated); Results first posted 2023-10-11 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2023-09

CONDITIONS: Oligometastatic Disease
Keywords: Oligo mets; Radiosurgery; Stereotactic Body Radiotherapy (SBRT) (Stereotactic radiosurgery (SRS) plus stereotactic radiotherapy (SRT))
MeSH Terms: conditions — Snyder Robinson syndrome | interventions — Radiosurgery; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Stereotactic Body Radiotherapy (SBRT) with/without chemotherapy (Experimental): Sequence of therapy: SRS/SBRT will be used for all sites of metastatic disease in close approximation to initiation of treatment for the primary disease site (within 6 weeks). Ideally, SRS/SBRT would occur first followed by treatment to primary site. However, in some circumstances surgical resection of the primary site could precede SRS/SBRT, especially if surgical resection is required for pathological confirmation of disease.
  Chemotherapy choice of agents is at the discretion of the treating medical oncologist; chemotherapy may be initiated after stereotactic radiosurgery treatment of the primary disease site has been completed.
  Interventions: Radiation: Stereotactic Radiosurgery (SRS); Drug: Chemotherapy

INTERVENTIONS:
Radiation: Stereotactic Radiosurgery (SRS) — Dose and fractionation will be dependent on the lesion location and lesion size, the exact fractionation and dose is at the discretion of the treating physician. A minimum of 48 hours must be used in between SRS treatments at each site. Patients may have SRS everyday or multiple SRS sessions in one day as long as the minimum time for each treatment site is met.
  Other Names: CyberKnife; Trilogy; True Beam
Drug: Chemotherapy — Chemotherapy choice of agents is at the discretion of the treating medical oncologist.

SUMMARY:
This study will evaluate the feasibility of radiosurgery for all metastatic sites in patients presenting with oligometastatic disease, defined here as 5 or fewer sites of metastatic disease involving 3 or fewer organ systems.

DETAILED DESCRIPTION:
Death from metastatic cancer is a common cause of death, accounting for 80-90% of cancer deaths. The classic thought process is that metastatic disease represents the continuum such that known metastatic disease is an inevitable harbinger for subsequent metastatic disease. However, it has been reported that a subset of patients with limited volume metastatic disease may have a better prognosis if given aggressive therapy. This group of patients has become known as "oligometastatic". These patients are potentially curable with stereotactic radiosurgery (SRS) or stereotactic radiotherapy (SRT) (collectively referred to as stereotactic body radiotherapy or SBRT) to the metastatic disease sites in combination with standard curative therapy to the primary site. Patients in this study receive SRS/SBRT to all sites of oligometastatic disease.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically (histologically or cytologically) proven diagnosis of solid malignancy within 8 weeks of registration
2. Eligible disease sites include the following

   * Breast
   * Prostate
   * GI (including colorectal, anal, esophagus, pancreas, gastric with the exception of colon cancer with resectable liver-only lesions)
   * Head and neck
   * Skin (melanoma and squamous cell carcinoma)
   * Lung (both small cell and non-small cell)
   * Sarcoma (both soft tissue and bone)
   * Gynecologic (endometrial, cervical, ovarian, vaginal, vulvar)
3. Patients are stage IV (M1) with any combination of T and N with oligometastatic disease as defined by 5 or fewer total sites of metastatic disease involving 3 or fewer organ systems

1 Examples of patients eligible for trial

* T3N2M1 NSCLC with 1 CNS metastatic lesion, 2 liver lesions, and 1 adrenal lesion.
* T4N1M1 colorectal cancer with 1 liver lesion, 4 bone lesions
* T3N0M1 gastric cancer with 1 supraclavicular lymph node, 2 liver lesions, and 2 CNS lesions 4Metastatic disease sites must be treatable with SRS (at discretion of treating physician).

  5Primary disease site must be able to be treated with curative intent 6Zubrod Performance Status 0-1 7Age ≥ 18 8CBC/differential obtained within 4 weeks prior to registration on study, with adequate bone marrow function defined as follows:
* Absolute neutrophil count (ANC) ≥ 1,800 cells/mm3;
* Platelets ≥ 100,000 cells/mm3;
* Hemoglobin ≥ 8.0 g/dl (Note: The use of transfusion or other intervention to achieve Hgb ≥ 8.0 g/dl is acceptable.); 9Women of childbearing potential and male participants must practice adequate contraception 10Patient must provide study specific informed consent prior to study entry.

Exclusion Criteria:

1. Ineligible disease sites include the following

   * Lymphoma
   * Leukemia
   * Multiple myeloma
   * Primary CNS
   * Peritoneal carcinomatosis
   * Colon cancer with resectable liver-only lesions
2. Examples of patients ineligible for trial

   * T1N1M1 NSCLC with 1 CNS lesion, 1 bone lesion, 1 adrenal lesion and a cervical lymph node (4 sites of metastatic disease)
   * T2N1M1 Gastric cancer with 6 liver lesions (more than 5 sites of metastatic disease)
3. Other

   * Lung cancer with pleural effusion (wet IIIB) are not eligible
   * Recurrent cancers are not eligible
   * Diffuse metastatic spread confined to one organ system is ineligible; examples of this include leptomeningeal spread in the CNS and peritoneal carcinomatosis.
4. Prior systemic chemotherapy for the study cancer; note that prior chemotherapy for a different cancer is allowable but cannot have any other primary cancer diagnosed or treated within the last 3 years other than cutaneous skin cancers. Patient may have previous chemotherapy as treatment of this previous malignancy as long as the chemotherapy has completed more than 3 years ago.
5. Prior radiotherapy to the region of the study cancer that would result in overlap of radiation therapy fields
6. Severe, active co-morbidity, defined as follows:

   * Unstable angina and/or congestive heart failure requiring hospitalization within the last 6 months;
   * Transmural myocardial infarction within the last 6 months;
   * Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration;
   * Hepatic insufficiency resulting in clinical jaundice and/or coagulation defects; note, however, that laboratory tests for liver function and coagulation parameters are not required for entry into this protocol.
   * Immuno-compromised patients.
7. Pregnancy or women of childbearing potential and men who are sexually active and not willing/able to use medically acceptable forms of contraception; this exclusion is necessary because the treatment involved in this study may be significantly teratogenic.
8. Oligometastatic disease sites not eligible based on concern for toxicity:

   * trachea involvement (direct invasion, tumors close to or abutting trachea are eligible)
   * heart (direct invasion or involvement, pericardial lymph nodes can be treated)
9. Patients unable to have an FDG-PET/CT scan, either through insurance coverage, patient decision or other reason are not eligible for this study.
10. Patients unable to have SRS through insurance coverage or ability to pay for SRS

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2013-06-07 (Actual); Primary Completion 2022-05-03 (Actual); Study Completion 2022-10-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steve J Burton, MD, Principal Investigator — UPMC Hillman Cancer Center
Locations (1):
- UPMC Hillman Cancer Center - Radiation Oncology, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Stereotactic Body Radiotherapy (SBRT) With/Without Chemotherapy: Sequence of therapy: SRS/SBRT will be used for all sites of metastatic disease in close approximation to initiation of treatment for the primary disease site (within 6 weeks). Ideally, SRS/SBRT would occur first followed by treatment to primary site. However, in some circumstances surgical resection of the primary site could precede SRS/SBRT, especially if surgical resection is required for pathological confirmation of disease.
  Chemotherapy choice of agents is at the discretion of the treating medical oncologist; chemotherapy may be initiated after stereotactic radiosurgery treatment of the primary disease site has been completed.
  Stereotactic Radiosurgery (SRS): Dose and fractionation will be dependent on the lesion location and lesion size, the exact fractionation and dose is at the discretion of the treating physician. A minimum of 48 hours must be used in between SRS treatments at each site. Patients may have SRS everyday or multiple SRS sessions in one day as long as the minimum time for each treatment site is met.
  Chemotherapy: Chemotherapy choice of agents is at the discretion of the treating medical oncologist.
Period: Overall Study
Arm/Group | Stereotactic Body Radiotherapy (SBRT) With/Without Chemotherapy
Started | 24
Completed | 24
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All patients enrolled in the study.
Arm/Group | Stereotactic Body Radiotherapy (SBRT) With/Without Chemotherapy
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.8333 (9.6534142)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 23
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 23
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Acceptable Toxicity of SRS/SBRT
Description: Number of distinct patients with toxicities of Grade 3 or less per CTCAE v4.0
Time Frame: Up to 3 Years (per patient)
Population: All treated patients able to be evaluated for toxicity grading.
Measure: Number; unit: participants
Arm/Group | Stereotactic Body Radiotherapy (SBRT) With/Without Chemotherapy
Number analyzed (Participants) | 2
participants
  GASTROINTESTINAL DISORDERS - Constipation : Grade 2 | 1
  GASTROINTESTINAL DISORDERS - Constipation : Grade 3 | 0
  GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS - Fatigue : Grade 2 | 1
  GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS - Fatigue : Grade 3 | 0
  METABOLISM AND NUTRITION DISORDERS - Anorexia : Grade 2 | 1
  METABOLISM AND NUTRITION DISORDERS - Anorexia : Grade 3 | 0
  MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDERS - Flank pain : Grade 2 | 0
  MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDERS - Flank pain : Grade 3 | 1
  MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDERS - Neck pain : Grade 2 | 1
  MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDERS - Neck pain : Grade 3 | 0
  VASCULAR DISORDERS - Hypertension : Grade 2 | 0
  VASCULAR DISORDERS - Hypertension : Grade 3 | 1

2. Primary Outcome: Presence of Multiple Metastatic Sites
Description: The presence of multiple metastatic disease sites (between 2 and 5 sites).
Time Frame: Up to 3 years (per patient)
Population: No data collected in the analysis population.
Arm/Group | Stereotactic Body Radiotherapy (SBRT) With/Without Chemotherapy
Number analyzed (Participants) | 0

3. Secondary Outcome: The Functional Assessment of Cancer Therapy - General (FACT-G) Quality of Life Score
Description: The Functional Assessment of Cancer Therapy - General (FACT-G) Quality of life Assessment is a patient self-administered 27-item questionnaire that measures health state in cancer patients in prior 7 days, including physical (PW), social (SW), emotional (EW), and functional (FW) well-being. Scoring: Five-point scale for each of the subscales is: 0 (not at all) to 4 (very much). PW has a Score range from 0-28. SW has a Score range from 0-28. EW has a Score range from 0-24. FW has a Score range from 0-28. Total overall score is thus from minimum of 0 to maximum of 108. Questions are phrased so that higher numbers indicate a better health state, leading to some items being reverse-scored.
Time Frame: At pre-treatment
Population: Participants that completed both pre and post treatment patient outcomes assessments.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stereotactic Body Radiotherapy (SBRT) With/Without Chemotherapy
Number analyzed (Participants) | 11
score on a scale
  Physical Well-being | 22.2727273 (4.5186482)
  Social Well-being | 25.4848485 (3.7693386)
  Emotional Well-being | 19.4545455 (3.2051096)
  Functional Well-being | 19.3636364 (6.3130457)
  Total Well-being | 86.5757273 (14.4845869)

4. Secondary Outcome: The Functional Assessment of Cancer Therapy - General (FACT-G) Quality of Score
Description: as for outcome 3
Time Frame: At post-treatment
Population: Participants that completed both pre and post treatment patient outcomes assessments.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stereotactic Body Radiotherapy (SBRT) With/Without Chemotherapy
Number analyzed (Participants) | 11
score on a scale
  Physical Well-being | 22.1282000 (4.5186482)
  Social Well-being | 24.0035692 (3.0955351)
  Emotional Well-being | 19.6250000 (4.3951633)
  Functional Well-being | 18.0651094 (7.0332731)
  Total Well-being | 83.7614375 (15.2425018)

5. Secondary Outcome: Local Control of Metastatic Disease
Description: Proportion of patients with local Complete Response (CR), Partial Response (PR) or Stable Disease (SD) after trial therapy as measured according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 at sites of metastatic disease. Per RECIST: (CR): Disappearance of all target lesions; (PR): At least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD. (SD) Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum LD since the treatment started.
Time Frame: Up to 5 years (per patient)
Population: No data collected in the analysis population
Arm/Group | Stereotactic Body Radiotherapy (SBRT) With/Without Chemotherapy
Number analyzed (Participants) | 0

6. Secondary Outcome: Local Control of Primary Disease
Description: Proportion of patients with local Complete Response (CR), Partial Response (PR) or Stable Disease (SD) after trial therapy as measured according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 at primary disease sites. Per RECIST: (CR): Disappearance of all target lesions; (PR): At least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD. (SD) Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum LD since the treatment started.
Time Frame: Up to 5 years
Population: No data collected in the analysis population.
Arm/Group | Stereotactic Body Radiotherapy (SBRT) With/Without Chemotherapy
Number analyzed (Participants) | 0

7. Secondary Outcome: Analysis of Patterns of Failure Post-SRS/SBRT
Description: The number of patients that experience oligometastatic disease progression/recurrence after treatment for their primary disease according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 at primary disease sites. Per RECIST, Progressive Disease (PD) includes the appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions.
Time Frame: Up to 5 years (per patient)
Population: Patients that received study treatment and were radiologically evaluated for confirmed disease progression.
Measure: Count of Participants; unit: Participants
Arm/Group | Stereotactic Body Radiotherapy (SBRT) With/Without Chemotherapy
Number analyzed (Participants) | 23
Participants | 18

8. Secondary Outcome: Two-year Overall Survival
Description: Percentage of participants alive at 2 years post start of treatment.
Time Frame: At 2 years (cohort)
Population: Participants that received study treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Stereotactic Body Radiotherapy (SBRT) With/Without Chemotherapy
Number analyzed (Participants) | 21
percentage of participants | 57.14

9. Secondary Outcome: Overall Survival (OS)
Description: Mean number of months patients remain alive from the day of trial enrollment until either an death from any cause or last follow-up.
Time Frame: Up to 5 years (cohort)
Population: Participants that received study treatment.
Measure: Mean (Standard Error); unit: months
Arm/Group | Stereotactic Body Radiotherapy (SBRT) With/Without Chemotherapy
Number analyzed (Participants) | 21
months | 32.7667 (5.1554)

ADVERSE EVENTS:
Time Frame: Adverse Events data were collected for up to 3 years per patient, and up to 9 years for the study population.
Description: Adverse Events were defined using National Cancer Institute (NCI) CTCAE version 4
Arm/Group | Stereotactic Body Radiotherapy (SBRT) With/Without Chemotherapy
All-Cause Mortality (participants affected / at risk) | 15/24
Serious Adverse Events (participants affected / at risk) | 1/24
Other Adverse Events (participants affected / at risk) | 2/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Stereotactic Body Radiotherapy (SBRT) With/Without Chemotherapy (N=24)
Cardiac Arrest (Cardiac disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Stereotactic Body Radiotherapy (SBRT) With/Without Chemotherapy (N=24)
Constipation (Gastrointestinal disorders) | 1
Coronary artery disease (Cardiac disorders) | 1
Fatigue (General disorders) | 1
Diabetes (General disorders) | 1
Hyperlipidemia (Investigations) | 2
Anorexia (Metabolism and nutrition disorders) | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Depression (Psychiatric disorders) | 1
Hypertension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-02-13): https://cdn.clinicaltrials.gov/large-docs/39/NCT01345539/Prot_SAP_000.pdf